CLINICAL TRIAL: NCT07205809
Title: In Vitro Comparison of Leakage in Endodontically Treated Teeth Obturated With Different Types of GP Coatings Using Bioceramic Sealer: A Randomized Controlled Trial.
Brief Title: Comparison of Leakage in Endodontically Treated Teeth Obturated With Different Types of Gutta Percha Coatings and Bioceramic Sealer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, Amna Amir, Principal Investigator, Pakistan Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SOD/ERB/2025/71
Record Dates: First submitted 2025-09-26; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Leakage Testing
Keywords: leakage; gutta percha; bioceramic; sealer
MeSH Terms: interventions — Gutta-Percha

STUDY DESIGN:
Intervention Model Description: This will be an in vitro experimental study conducted on extracted human teeth. A total of 60 single-rooted teeth will be collected according to inclusion and exclusion criteria. Using a non-probability consecutive sampling technique, the teeth will be instrumented with ProTaper NEXT files up to size F3 and then divided into two groups (n=30 each). Group 1 will be obturated with bioceramic sealer and bioceramic-coated gutta-percha, while Group 2 will be obturated with bioceramic sealer and conventional gutta-percha. Microleakage will be evaluated in millimeters and the data analyzed using SPSS (version 25). This model allows for controlled comparison of sealing ability between the two obturation techniques.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I: Bioceramic sealer + Bioceramic coated GP) (Experimental): Extracted single-rooted teeth obturated with bioceramic-coated gutta-percha in combination with a bioceramic sealer. This arm evaluates the sealing ability of the newer coated obturation material.
  Interventions: Procedure: bioceramic coated gutta percha
- Group II (Bioceramic sealer + conventional (non-coated) GP) (Active Comparator): Extracted single-rooted teeth obturated with conventional (non-coated) gutta-percha in combination with a bioceramic sealer. This arm serves as the reference/control to compare sealing ability against the experimental mate
  Interventions: Procedure: conventional(non-coated) gutta percha

INTERVENTIONS:
Procedure: bioceramic coated gutta percha — Experimental Arm (Bioceramic-coated GP + Bioceramic Sealer):
  Specimens will be obturated using bioceramic-coated gutta-percha cones in combination with bioceramic sealer after canal preparation with ProTaper NEXT files up to size F3.
  Arms: Group I: Bioceramic sealer + Bioceramic coated GP)
Procedure: conventional(non-coated) gutta percha — Active Comparator Arm (Conventional GP + Bioceramic Sealer):
  Specimens will be obturated using conventional (non-coated) gutta-percha cones in combination with the same bioceramic sealer after canal preparation with ProTaper NEXT files up to size F3.
  Arms: Group II (Bioceramic sealer + conventional (non-coated) GP)

SUMMARY:
In vitro study to compare the sealing ability of bioceramic-coated gutta-percha with bioceramic sealer against conventional gutta-percha with bioceramic sealer in root canal obturation. A total of 60 extracted human single-canal teeth will be prepared and obturated according to standardized protocols, then evaluated for microleakage. Data will be analyzed using SPSS (version 25) with appropriate non-parametric tests at a significance level of p<0.05. The outcomes are expected to identify the more effective obturation material combination in achieving a fluid-tight seal, thereby contributing to improved success rates in endodontic therapy.

DETAILED DESCRIPTION:
This study will evaluate the sealing ability of bioceramic-coated gutta-percha compared with conventional gutta-percha, both used in combination with a bioceramic sealer, in single-rooted teeth. A total of 60 extracted human teeth will be prepared and divided into two groups for obturation.

A total of 60 single-canal, extracted human teeth will be selected according to inclusion and exclusion criteria through non-probability consecutive sampling. The teeth will be cleaned and shaped using ProTaper NEXT endodontic files (DENTSPLY Tulsa Dental Specialties, DENTSPLY International, Inc., USA) to size F3, then specimens will be randomly divided into two groups (n=30 each) using the lottery method.

Group I: Bioceramic sealer + Bioceramic coated GP Group II: Bioceramic sealer + conventional (non-coated) GP

Obturation will be done using the cold lateral condensation technique. All specimens will be soaked in 1% Methylene Blue dye at 37°C for seven days. Afterward, roots will be grounded (longitudinally) mesiodistally with abrasive paper or diamond slit until gutta percha and dye visible both coronally and apically. Images of each root will be taken using a digital camera (DSLR), including a mm ruler and the number label. Image J software will measure the maximum linear dye penetration (in millimeters) along the coronal and apical boundaries of teeth.

The data will be entered and analyzed using the Statistical Package for Social Sciences (SPSS, version 25). Descriptive statistics (mean ± SD) will be calculated. Differences in leakage (in mm) between the two groups will be assessed using the Kruskal-Wallis test. If significant, pairwise comparisons will be performed using the Mann-Whitney U test with Bonferroni correction. A p-value < 0.05 will be considered statistically significant. Results will be presented in tabular form.

Microleakage will be measured and statistically analyzed to determine the more effective material combination for achieving a fluid-tight seal in root canal therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Extracted human teeth with single canal and mature root apex

Exclusion Criteria:

1. Teeth with calcified (non-negotiable) canals.
2. Teeth with internal/external root resorption (as seen on radiograph)
3. Teeth with caries extending to the floor of pulp chamber.
4. Teeth with a single canal but open apex.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-05 (Estimated); Primary Completion 2026-05-05 (Estimated); Study Completion 2026-06-12 (Estimated)

PRIMARY OUTCOMES:
post obturation leakage | six months
  assessment of leakage in obturated teeth in experimental group and control group via dye penetration method. specimens soaked in 1% methylene blue dye for seven days

CONTACTS AND LOCATIONS:
Overall Officials: Amna Amir, BDS, Principal Investigator — School of Dentistry, Shaheed Zulfiqar Ali Bhutto Medical University, Islamabad.
Locations (1):
- School of Dentistry, Shaheed Zulfiqar Ali Bhutto Medical University, Islamabad, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No